CLINICAL TRIAL: NCT04150601
Title: Evaluation of SIMEOX Technology on Volumes and Flows Generated in Healthy Subjects and Patients With COPD
Brief Title: Effects of SIMEOX on Flow and Volume in Healthy Subjects and Patients With COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Principal Investigator, William Poncin, PT, PhD, Principal Investigator, Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SIMEOX-002
Record Dates: First submitted 2019-10-31; First posted 2019-11-05 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Healthy; Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Spontaneous slow vital capacity (Active Comparator): Participants will have to perform a slow vital capacity according to the guidelines, from total lung capacity to residual volume
  Interventions: Other: Spontaneous Exhalation
- SIMEOX (Active Comparator): Participants will have to perform a passive exhalation using the SIMEOX, starting from total lung capacity and going until achieving residual volume
  Interventions: Device: SIMEOX
- PEP (Active Comparator): Participants will have to perform an active exhalation using a PEP device, starting from total lung capacity and going until achieving residual volume
  Interventions: Device: PEP

INTERVENTIONS:
Device: SIMEOX — SIMEOX is a device generating a succession of gentle depression at the mouth.
  Arms: SIMEOX
Device: PEP — A PEP device (Pari-PEP) will be used to provoke a positive expiratory pressure while exhaling, thereby stabilizing the airways during expiration.
  Arms: PEP
Other: Spontaneous Exhalation — A slow vital capacity maneuver will be performed according to the guidelines, from total lung capacity to residual volume
  Arms: Spontaneous slow vital capacity

SUMMARY:
This study will investigate the effects on the SIMEOX technology on flow and volume generated in healthy subjects and patients with COPD

DETAILED DESCRIPTION:
This is a crossover study assessing the immediate physiological effects of SIMEOX and a PEP device on the exhalation phase in healthy subjects and patients with COPD.

Participants will perform (1) a slow vital capacity, (2) a maximal expiration from total lung capacity to residual volume with SIMEOX, (3) a maximal expiration from total lung capacity to residual volume with a PEP device.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects: able to understand the instructions, no acute or chronic respiratory upper or lower airway disease, normal lung function.
* Patients with COPD: able to understand the instructions; FEV1<80% predicted value, naive to the SIMEOX device.

Exclusion Criteria:

* Healthy subjects: obesity (BMI > 30kg/m²); active or former smoker; severe scoliosis; cardiovascular or neuromuscular disease.
* Patients with COPD: obesity (BMI > 30kg/m²); severe scoliosis; cardiovascular or neuromuscular disease.

Ages: 45 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-11-16 (Actual); Study Completion 2021-11-16 (Actual)

PRIMARY OUTCOMES:
Change in expiratory volume | 5 minutes
  Expiratory volume change between the 3 conditions (spontaneous expiration, SIMEOX and PEP).
Change in expiratory flow | 5 minutes
  Expiratory flow change between the 3 conditions (spontaneous expiration, SIMEOX and PEP).

CONTACTS AND LOCATIONS:
Locations (1):
- Cliniques universitaires Saint-Luc, Brussels, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: No